CLINICAL TRIAL: NCT02727764
Title: A Single Dose Clinical Trial to Study the Safety of ART-I02 in Patients With Arthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arthrogen (Industry)
Collaborators: Centre for Human Drug Research (CHDR) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-I02-001-NL
Record Dates: First submitted 2016-03-09; First posted 2016-04-05 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-02

CONDITIONS: Arthritis, Rheumatoid; Osteo Arthritis
Keywords: Arthritis; Gene therapy; Phase Ib; Intra-articular
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort I (Experimental): ART-I02 1.2x10e12 vg/ CMC joint, 1.2x10e12 vg/ MCP joint, 0.6x10e12 vg/ PIP joint or 0.3x10e12 vg/ DIP joint single intra-articular injection
  Interventions: Genetic: ART-I02
- Cohort II (Experimental): ART-I02 1.2x10e12 vg/ CMC joint, 1.2x10e13 vg/ MCP joint, 0.6x10e13 vg/ PIP joint or 0.3x10e13 vg/ DIP joint single intra-articular injection
  Interventions: Genetic: ART-I02
- Cohort III (Experimental): ART-I02 1.2x10e12 vg/ CMC joint, 1.2x10e13 vg/ MCP joint, 0.6x10e13 vg/ PIP joint or 0.3x10e13 vg/ DIP joint ART-I02 or maximum Tolerated Dose (MTD) as assessed in cohorts I and II: single intra-articular injection
  Interventions: Genetic: ART-I02

INTERVENTIONS:
Genetic: ART-I02 — Single Intra-articular injection in the carpometacarpal (CMC), metacarpophalangeal (MCP), proximal interphalangeal (PIP), or distal interphalangeal (DIP) joint
  Other Names: Recombinant AAV type2/5 containing a hIFN-b gene

SUMMARY:
This study will evaluate the safety and tolerability of a single intra-articular administration of ART-I02 (AAV5.NF-kB.IFN-β), a recombinant adeno-associated virus (AAV) type 2/5 vector in subjects with Rheumatoid Arthritis (RA) or Osteoarthritis (OA) and active arthritis of the carpometacarpal (CMC), metacarpophalangeal (MCP), proximal interphalangeal (PIP), or distal interphalangeal (DIP) joints.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic, chronic, inflammatory disorder leading to accelerated joint inflammation causing pain, swelling and limited motion of joints, ultimately leading to the development of joint destruction and deformity in the majority of patients. Virtually all peripheral joints can be affected by RA, although the most commonly affected joints are those of wrists, hands, knees, and feet.

During the last decade, treatment with biologicals (e.g. TNF-inhibitors), together with improved timing and dosing of conventional therapy, has significantly improved the outcome in a significant proportion of RA patients. The advent of biologicals and implementation of more intensive treatment protocols has significantly improved the outcome in a significant proportion of RA patients and prevented disabilities. However, drug-free remissions are still rare and hence most RA patients require continued immunosuppressive treatment which predisposes them to potentially serious infections.

Also up to 50% of RA patients continue to suffer from symptomatic disease. Intra-articular glucocorticoids are often used in these patients, e.g. when single joints are inflamed. The duration of their effect is however variable. It regularly occurs in clinical practice that reasonable clinical remission in rheumatoid arthritis patients is achieved with current treatment options, but that one or more joints still display persistent signs of inflammation while the inflammation of other joints has been greatly reduced. This means that for the joint(s) still affected by active inflammation other therapies are required.

There is thus a large unmet need for additional RA therapies with good tolerability and efficacy profiles that can be used in patients who are not eligible for standard treatment, and in those who despite standard treatment suffer from inflamed joints. Local gene therapy with IFN-β could be a potential treatment to fulfil this unmet need; the selection of IFN-β as the therapeutic protein is based on the notion that IFN-β has anti-inflammatory, bone and cartilage protective effects, which have been extensively demonstrated in non-clinical studies.

Osteoarthritis (OA) is a multifactorial joint disease that involves degeneration of articular cartilage, causing pain, limited range of motion of joints and thereby disability. Although aetiology is largely unknown, important factors such as genetic pre-disposition, mechanical and biochemical stress are known to play a role in this multi factorial disease. Ligaments, menisci, and muscles can also be affected, and osteophytes may develop, causing additional pain.

Current treatment options of OA are restricted to symptomatic treatment to mitigate pain, rather than proactively preventing progression of disease. These treatment options in early stage OA consist of non-pharmacological therapies, such as advice in joint strain in periods of complaints, which can potentially be aided by splint therapy and targeted exercises. In a later stage of OA, systemic or local topically applied analgesics are commonly utilized. Another option is the injection of compounds in the joints, but neither corticosteroids nor hyaluronic acid injections have proven to significantly improve pain compared to placebo. Surgical options in hand OA exist, but are only recommended in patients with severe motion restriction and these surgeries may not be beneficial to all patients Although there are a number of options aiding patients with OA, currently there are less treatment options for osteoarthritis (OA) than for RA and most focus on mitigation of pain. In both RA and OA, this means that for the joint(s) still affected by active inflammation other therapies are required.

ART-I02 is an investigational new drug, expressing human IFN-β from a recombinant (r) adeno-associated virus type 5 (rAAV5) β under the influence of a promoter, which is induced by an inflammatory stimulus. Due to the relapsing nature of RA, therapeutic expression should be maximal during flare-ups of the disease. This is achieved by employing the NF-kB responsive promotor to regulate expression of IFN-β. Under inflammatory conditions, the NF-kB responsive promoter will be activated in the synovium and will upregulate the expression of hIFN-β and turned down during remission. In this way, transgene expression can be controlled, following the intermittent course of disease.

In this phase I open label, dose escalating study the safety of a single intra-articular ART-I02 injection in patients with RA or OA and active arthritis of the metacarpophalangeal (MCP), proximal interphalangeal (PIP), or distal interphalangeal (DIP) joint with an indication for surgical intervention which includes removal of the synovium. In a two-phase staggered dose escalation design, dosing will start with a low dose (1.2x1012 vg/ MCP joint, 0.6x1012 vg/ PIP joint or 0.3x1012 vg/ DIP joint) and progress to the highest dose of 1.2x1013 vg/ MCP joint, 0.6x1013 vg/ PIP joint or 0.3x1013 vg/ DIP joint. Three patients will be enrolled at each of the two dose levels. Enrolment of a subject within each of the two cohorts will not proceed until the safety data through day 7 from the previous subject have been reviewed/evaluated by the investigator. After dosing of the last subject in cohort I and II, a dosing pause of two weeks is included to allow an assessment of the safety data by the Data Review Committee. All available safety data including a minimum of 2 weeks of data (safety and tolerability data through day 14 post ART-I02 administration) from the 3rd patient of cohort I and II (medical history, vital signs, physical examination, laboratory parameters, ECG and adverse events) will be reviewed. Only after a thorough assessment of these safety data enrolment in the next cohort will continue.

In cohort III six patients will be administered the highest safety dose of ART-I02 as determined in the previous dose escalating cohorts (cohorts I and II). Cohort III is added to the study to substantiate the safety profile of the highest tolerated dose of ART-I02.

Subjects will be followed for 24 weeks after the single intra-articular injection of ART-I02 for safety. Although the study is not designed to demonstrate a clinical effect, (clinical) efficacy parameters will be evaluated. After this period subjects will be included in a long term follow-up study for another 4.5 years to assess long term safety.

The consideration to treat one joint in this clinical study is that it provides the opportunity to examine the administration of a single dose at the site where the promoter is activated and where the therapeutic protein IFN-β is required. Patients who have an indication for a surgical intervention for the affected target joint will be recruited for this study. With this approach a possible benefit for the patients can be obtained (postponing the surgical intervention), while at the same time it provides the opportunity to mitigate risk caused by untoward effects due to persistence of the vector (planned surgical intervention will be carried out earlier).

ELIGIBILITY:
Inclusion criteria

1. Patients ≥18 years of age.
2. Patient have to be diagnosed with RA according to the 2010 American College of Rheumatology/ European league against rheumatism (ACR/EULAR) criteria for the classification of RA, outlined in appendix B or OA as confirmed by their treating physician/specialist.
3. Patient is scheduled for surgical intervention of the target joint.
4. Inflammation of the CMC, MCP, PIP or DIP joint as confirmed by MRI.
5. Written informed consent, able and willing to comply with the requirements of the study protocol.
6. Judged to be in general good health with, in the opinion of the investigator, no other clinically significant and relevant abnormalities of medical history, and no abnormalities at the physical examination, vital signs, electrocardiography (ECG) and laboratory safety tests, performed at the screening visit and/or prior to administration of ART-I02.
7. Females are not pregnant nor lactating. All patients use effective contraception in combination with barrier contraception for the first three months after administration or until three consecutive semen samples are negative.

Exclusion criteria

1. Arthrodesis or joint replacement of the target CMC, MCP, PIP or DIP joint prior to inclusion.
2. Known hypersensitivity to natural or recombinant hIFN-β, or to any excipients.
3. Contra-indication for intra-articular treatment.
4. Presence of neutralising antibody (Nab) titers against adeno-associated virus type 5 (AAV5) and/or hIFN-β.
5. Active infectious disease of any nature, including clinical active viral infections.
6. Previous treatment with an AAV-5 vector.
7. Poor functional status, defined as being bed-bound.
8. Participation in an investigational drug or device study within 90 days prior to screening or more than 4 times per year.
9. Positive for human immunodeficiency virus (HIV) infection, hepatitis C antibodies or hepatitis B surface antigen.
10. Positive for anti-double-stranded DNA antibodies (dsDNA).
11. History of liver function abnormality requiring treatment, drug induced liver injury, chronic liver disease, excessive alcohol consumption or chronic alcohol induced disease.
12. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN), or bilirubin > 2 x ULN. If a patient has AST or ALT > 2 x ULN but < 2.5 x ULN, re-assessment is allowed at the investigator's discretion.
13. Severely impaired renal function (estimated glomerular filtration rate ≤ 30 mL/min according to the Cockcroft-Gault formula).
14. Patient donated or lost approximately 500 ml blood within 4 months prior to the screening visit
15. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude
16. Serious medical disease, such as severe liver or kidney disease, uncompensated congestive heart failure, myocardial infarction within six months, unstable angina, uncontrolled hypertension, severe pulmonary disease or active asthma, demyelinating neurological disease, depression or a history of depression, history of seizures or epilepsy, uncontrolled epilepsy, or history of cancer (other than cutaneous basal and squamous cell carcinoma or cervical intraepithelial neoplasia) with less than five years documentation of a disease-free state, recurrent opportunistic infections or other concurrent medical condition that, in the opinion of the investigator, would make the patient unsuitable for the study.
17. Investigator has concerns regarding the safe participation of the patient in the trial or for any other reasons: the investigator considers the patient inappropriate for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent (serious) adverse events | Five years
  Treatment emergent (serious) adverse events

SECONDARY OUTCOMES:
Change from baseline for clinical signs and symptoms of the target joint evaluated by the Composite Change Index (CCI) at week 1, week 2, week 4, week 8, week 12, week 16, week 20 and week 24 post administration of ART-I02. | Baseline, week 1, week 2 , week 4, week 8, week 12, week 16, week 20 and week 24 post administration of ART-I02
  Change from baseline of clinical signs and symptoms as measured by the aggregate score of the individual components of the CCI. Calculation of the CCI is based on changes of its components from baseline. The total CCI ranges from 0 (no effect or deterioration) to 10 (maximal effect). Successful treatment is defined as CCI ≥5.
Change from baseline on synovitis and osteitis in the injected joint (target joint) evaluated by Magnetic Resonance Imaging (MRI) 12 and 24 weeks after administration of ART-I02 using the OMERACT RA MRI scoring system (RAMRIS). | 12 and 24 weeks after administration of ART-I02
  Change from baseline on synovitis and osteitis will be assessed by evaluating the aggregate scores of the components of the RAMRIS scoring system at week 12 and week 24. Synovitis will be assessed in three wrist regions (distal radioulnar joint, radiocarpal joint, intercarpal and carpometacarpal joints) and each MCP joint. Scale: 0-3 in increments of 33 % of the synovial compartment. Bone erosions will be assessed in each bone (wrists - carpal bones, distal radius, distal ulna, metacarpal bases; MCP joints - metacarpal heads, phalangeal heads) is scored separately . Scale: 0-10 in increments of 10 % of articular bone loss. Osteitis will be assessed by scoring each bone separately. Scale: 0-3 in increments of 33 % of bone oedema
Vector DNA in whole peripheral blood, semen, urine, feces, and saliva | Up to 24 weeks but maximally until such time that three consecutive samples have been tested negative
  To evaluate shedding of ART-I02 in blood, urine, faeces and saliva
Induction of humoral immune responses against AAV5 by measuring antibodies against AAV5 and neutralizing antibodies against AAV5 at baseline, week 4 and week 24 post administration | Baseline, week 4 and week 24 post administration
  To assess immune responses against adeno-associated virus serotype 5 (AAV5) after a single intra-articular dose of ART-I02
Induction of humoral immune responses against hIFN-β by measuring antibodies against IFN-β and neutralizing antibodies against hIFN-β at baseline, week 4 and week 24 post administration | Baseline, week 4 and week 24 post administration
  To assess immune responses against human interferon beta (hIFN-β) after a single intra-articular dose of ART-I02.
Induction of cellular immune responses against AAV5 by measuring T cell responses against AAV5 at baseline week 4, 8, 12, 16 and week 24 post administration | Baseline, week 4, 8, 12, 16 and week 24 post administration
  To assess T-cell response against AAV5
Induction of cellular immune responses against hIFN-β by measuring T cell responses against hIFN-β at baseline week 4, 8, 12, 16 and week 24 post administration | Baseline, week 4, 8, 12, 16 and week 24 post administration
  T-cell response against hIFN-β
Improvement of the target joint will be assessed by extension and flexion evaluation | Baseline, week 1, week 2, week 4, week 8, week 12, week 16, week 20 and week 24
  To explore the response to a single intra-articular dose of ART-I02 by assessing MCP, PIP, DIP extension/ flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Koos Burggraaf, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Centre for Human Drug Research (CHDR), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vrouwe JPM, Meulenberg JJM, Klarenbeek NB, Navas-Canete A, Reijnierse M, Ruiterkamp G, Bevaart L, Lamers RJ, Kloppenburg M, Nelissen RGHH, Huizinga TWJ, Burggraaf J, Kamerling IMC. Administration of an adeno-associated viral vector expressing interferon-beta in patients with inflammatory hand arthritis, results of a phase I/II study. Osteoarthritis Cartilage. 2022 Jan;30(1):52-60. doi: 10.1016/j.joca.2021.09.013. Epub 2021 Oct 6. PMID 34626797